CLINICAL TRIAL: NCT02617940
Title: Effectiveness of Sealants in Cavitated Enamel Lesions on Occlusal Surfaces of Primary and Permanent Molars in Children
Brief Title: Efficacy of Sealants in Cavitated Enamel Lesions on Occlusal Surfaces in Children
Acronym: SLM1661
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty Sao Leopoldo Mandic Campinas (Other)
Responsible Party: Principal Investigator, Jose Carlos P Imparato, PhD, Senior Lecturer, Faculty Sao Leopoldo Mandic Campinas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SLM1
Record Dates: First submitted 2015-11-22; First posted 2015-12-01 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Fissure Sealants; Oral Hygiene Orientation
Keywords: dental caries; primary tooth; resin-based sealants
MeSH Terms: conditions — Dental Caries | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fissure sealant (Experimental): single placement of resin-based sealant on occlusal surface and oral hygiene orientation
  Interventions: Other: fissure sealant
- oral hygiene orientation (Placebo Comparator): single application of water on occlusal surface and oral hygiene orientation
  Interventions: Other: oral hygiene orientation

INTERVENTIONS:
Other: fissure sealant — Surfaces allocated to this group will be treated with resin-based sealant (FluroShield®, Dentsply, United States of America) according to the manufacturer's instructions.
  Initially, local anesthesia and rubber dam adaptation will be performed. Then, 37% phosphoric acid will be applied on the surface for 30 seconds, followed by spray of water/air for at least 15 seconds. The sealant will be dispensed on the occlusal surface and light cured for 20 seconds (Optilight Max, Gnatus, Brazil).
  Arms: fissure sealant
Other: oral hygiene orientation — Surfaces allocated to this group will be treated with sterile water application, as a placebo, without anesthesia and rubber dam. The active treatment in this group will be only oral hygiene orientations.
  Arms: oral hygiene orientation

SUMMARY:
The aim of this study is to evaluate the efficacy of oral hygiene orientation singly, compared to resin-based sealants in controlling occlusal cavitated enamel lesions on primary and permanent molars. For this, 273 occlusal surfaces of primary molars and 273 occlusal surfaces of first permanent molars on 4-9 years-old children with an enamel cavitated lesion will be selected in 9 cities of Brazil. The surfaces will be randomly divides into 2 groups: oral hygiene orientation and resin-based sealant. The surfaces will be evaluated after 6 and 12 months regarding clinical and radiographic lesions progression. The costs and cost-efficacy of these treatments, children's discomfort, parents'/guardians' satisfaction and impact on quality of life will also be investigated. Poisson regression analysis will be performed in order to compare the groups, through clinical and radiographic criteria. This test will also be used to assess the association between the group and patient discomfort and parents' satisfaction. Time, costs and impact on quality of life of the treatments will be compared by Student's t test. For all analyses, the significance level will be set at 5%.

ELIGIBILITY:
Inclusion Criteria:

* parents or legal guardians accept and sign the informed consent form.
* children must have at least one molar with caries lesion classified as ICDAS active score 3.

Exclusion Criteria:

* children with special needs and/or systemic diseases with oral impairment.
* teeth with spontaneous painful symptoms or necrotized and teeth presenting restorations, sealants, cavitated caries lesions in dentin or other types of formation defects.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 546 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Sealants clinical efficacy | Every 6 months up to 12 months
  The clinical evaluation will be performed by one blinded examiner. If the surface is sealed, the examiner will classify it according to described by Pardi et al. (2005); if the surface is without material, the examiner will use the International Caries Detection and Assessment System (ICDAS) criteria (Ismail et al., 2007).
Sealants radiographic efficacy | Every 6 months up to 12 months
  The radiographic evaluation will be performed by two blinded examiners, which will evaluate the four patients' radiographies independently, two by two, without knowing the chronological order of them. The efficacy of the treatment will be related to the presence or absence of increasing radiolucent area. They will also classify each radiograph using Ekstrand criteria (Ekstrand et al., 1997) and analyze them in a software (ImageJ 1.49, National Institute of Health, United States of America) in order to make the radiographic subtraction.

SECONDARY OUTCOMES:
Sealants and oral hygiene orientation costs | Baseline
  Treatment costs will be calculated for each treatment technique considering professional costs and procedure costs. In order to calculate the professional cost, the time spent in each session will be converted in hours and multiplied by the medium income of the dentist per hour as related by the Brazilian Ministry of Labour and Employment. To estimate the procedure cost, it will be considered both variable cost, which includes electricity and equipment depreciation, and materials cost. To calculate the equipment depreciation (peripherals, dental chair and instrumental), we will consider their price, the lifespan of five years and a monthly use of 160 hours, resulting in an estimate value per hour. All materials used in each procedure will have their quantity registered. Prices will be inferences from the market value converted in US Dollars.
Sealants cost-efficacy | Through study completion (12 months)
  The costs of each treatment procedure will be calculated and compared with threshold values for intervention cost-effectiveness by region, determined by World Health Organization (http://www.who.int/choice/costs/CER_levels/en/).
Impact on children's quality of life of sealants or oral hygiene orientation | 6 and 12 months
  The oral health related to quality of life will be measured using a validated questionnaire according to the children's age. The Early Childhood Oral Health Impact Scale (ECOHIS) will be applied with 4-5 years old children and Child Perceptions Questionnaire will be used for 6-9 (CPQ8-10) years old children. They will be applied immediately before the procedure and on 6 months follow-up
Children self-reported discomfort | Baseline
  The discomfort of each type of treatment will be evaluated using the facial scale of Wong-Baker (Wong, Baker, 1998). This scale indicates the discomfort of an individual who has to choose among six faces. The first image is a smiling happy face, indicating no discomfort, followed by gradually less cheerful expressions, up to the last one which is a very sad face covered by tears, indicating great discomfort. The participant will be asked to choose the face that is more similar to how he/she felt during the treatment immediately after the procedure. This answer should be given solely by the child, which means no parental or professional interferences.
Parents' reported satisfaction with treatment | 6 months
  The parents'/guardians' satisfaction with treatment will be evaluated using a questionnaire. It will be applied only at the 6-months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jose CP Imparato, PhD, Principal Investigator — Faculty Sao Leopoldo Mandic Campinas
Locations (1):
- Jose Carlos Pettorossi Imparato, São Paulo, Brazil

REFERENCES:
- [Background] Erdemir U, Sancakli HS, Yaman BC, Ozel S, Yucel T, Yildiz E. Clinical comparison of a flowable composite and fissure sealant: a 24-month split-mouth, randomized, and controlled study. J Dent. 2014 Feb;42(2):149-57. doi: 10.1016/j.jdent.2013.11.015. Epub 2013 Dec 1. PMID 24296163
- [Background] Ahovuo-Saloranta A, Forss H, Walsh T, Hiiri A, Nordblad A, Makela M, Worthington HV. Sealants for preventing dental decay in the permanent teeth. Cochrane Database Syst Rev. 2013 Mar 28;(3):CD001830. doi: 10.1002/14651858.CD001830.pub4. PMID 23543512
- [Background] Morales-Chavez MC, Nualart-Grollmus ZC. Retention of a resin-based sealant and a glass ionomer used as a fissure sealant in children with special needs. J Clin Exp Dent. 2014 Dec 1;6(5):e551-5. doi: 10.4317/jced.51688. eCollection 2014 Dec. PMID 25674325
- [Background] Ricketts DN, Ekstrand KR, Martignon S, Ellwood R, Alatsaris M, Nugent Z. Accuracy and reproducibility of conventional radiographic assessment and subtraction radiography in detecting demineralization in occlusal surfaces. Caries Res. 2007;41(2):121-8. doi: 10.1159/000098045. PMID 17284913
- [Background] Hilgert LA, Leal SC, Mulder J, Creugers NH, Frencken JE. Caries-preventive Effect of Supervised Toothbrushing and Sealants. J Dent Res. 2015 Sep;94(9):1218-24. doi: 10.1177/0022034515592857. Epub 2015 Jun 26. PMID 26116491
- [Background] Schwendicke F, Jager AM, Paris S, Hsu LY, Tu YK. Treating pit-and-fissure caries: a systematic review and network meta-analysis. J Dent Res. 2015 Apr;94(4):522-33. doi: 10.1177/0022034515571184. Epub 2015 Feb 20. PMID 25710951
- [Background] Walsh T, Worthington HV, Glenny AM, Appelbe P, Marinho VC, Shi X. Fluoride toothpastes of different concentrations for preventing dental caries in children and adolescents. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD007868. doi: 10.1002/14651858.CD007868.pub2. PMID 20091655
- [Background] Guedes RS, Piovesan C, Floriano I, Emmanuelli B, Braga MM, Ekstrand KR, Ardenghi TM, Mendes FM. Risk of initial and moderate caries lesions in primary teeth to progress to dentine cavitation: a 2-year cohort study. Int J Paediatr Dent. 2016 Mar;26(2):116-24. doi: 10.1111/ipd.12166. Epub 2015 Apr 28. PMID 25923059
- [Background] Liu BY, Lo EC, Chu CH, Lin HC. Randomized trial on fluorides and sealants for fissure caries prevention. J Dent Res. 2012 Aug;91(8):753-8. doi: 10.1177/0022034512452278. Epub 2012 Jun 26. PMID 22736448
- [Background] Mendes FM, Braga MM. Caries detection in primary teeth is less challenging than in permanent teeth. Dent Hypotheses 4: 17-20, 2013.
- [Background] Martins-Junior PA, Vieira-Andrade RG, Correa-Faria P, Oliveira-Ferreira F, Marques LS, Ramos-Jorge ML. Impact of early childhood caries on the oral health-related quality of life of preschool children and their parents. Caries Res. 2013;47(3):211-8. doi: 10.1159/000345534. Epub 2012 Dec 13. PMID 23257929
- [Background] Barbosa Tde S, Gaviao MB. [Quality of life and oral health in children - Part II: Brazilian version of the Child Perceptions Questionnaire]. Cien Saude Colet. 2011 Jul;16(7):3267-76. doi: 10.1590/s1413-81232011000800026. Portuguese. PMID 21808914
- [Background] Wong DL, Baker CM. Smiling faces as anchor for pain intensity scales. Pain. 2001 Jan;89(2-3):295-300. doi: 10.1016/s0304-3959(00)00375-4. No abstract available. PMID 11291631
- [Background] Pardi V, Pereira AC, Ambrosano GM, Meneghim Mde C. Clinical evaluation of three different materials used as pit and fissure sealant: 24-months results. J Clin Pediatr Dent. 2005 Winter;29(2):133-7. doi: 10.17796/jcpd.29.2.e44h17387x324345. PMID 15719917
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Ekstrand KR, Ricketts DN, Kidd EA. Reproducibility and accuracy of three methods for assessment of demineralization depth of the occlusal surface: an in vitro examination. Caries Res. 1997;31(3):224-31. doi: 10.1159/000262404. PMID 9165195